CLINICAL TRIAL: NCT01603810
Title: An Investigation of the Correlation Between OCT and Histology in Defining the Margins of Periocular Basal Cell Carcinoma
Brief Title: Evaluating In Vivo OCT Imaging for Periocular Basal Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maidstone & Tunbridge Wells NHS Trust (Other)
Responsible Party: Principal Investigator, Henry Smith, Oculoplastics Fellow, Maidstone & Tunbridge Wells NHS Trust
Other Study IDs: MTW001
Record Dates: First submitted 2012-05-19; First posted 2012-05-22 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Basal Cell Carcinoma
Keywords: Basal cell carcinoma; Optical Coherence Tomography
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- BCC: Adult of any age or gender with capacity to give informed consent who has a basal cell carinoma requiring surgical excision and involving the periocular skin
  Interventions: Other: OCT

INTERVENTIONS:
Other: OCT — Optical coherence tomography of periocular basal cell carcinoma

SUMMARY:
Optical coherence tomography (OCT) is an imaging technique which shows the internal structure of living tissue (in vivo). It is safe, quick and painless to perform, and does not damage the tissue in any way. Recent advances in the technology mean that it can now be used to take images of the internal structure of the skin. This is useful because certain conditions, such as skin cancers, alter this structure. At present a suspected skin cancer is identified by taking a sample (a biopsy) which is analysed under the microscope to confirm the diagnosis. The cancer is then excised including a margin of apparently healthy-looking skin around it to ensure that the entirety of the tumour is removed. The excised tumour is then analysed again under a microscope to confirm that it was indeed completely removed (histology), after which a further operation is required to repair the defect.

The purpose of this study is to evaluate OCT imaging of a particular type of skin cancer called a basal cell carcinoma (BCC), and in particular BCCs affecting the skin around the eyes (periocular). The study will compare the ability of OCT to define the margin of the BCC with the current 'gold standard' of histology. OCT could potentially improve the investigators ability to define the margins of the tumour before surgery and become a guide for minimally invasive surgery. The preservation of healthy tissue represents a priority, particularly in the area of the skin surrounding the eye.

ELIGIBILITY:
Inclusion Criteria:

* Adults of any age or gender who have capacity to give informed consent, and who have periocular basal cell carcinoma requiring surgical excision

Exclusion Criteria:

* Children, vulnerable adults, inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with periocular basal cell carcinoma
Sampling Method: Non-Probability Sample

CONTACTS AND LOCATIONS:
Overall Officials: Henry B Smith, FRCOphth, Principal Investigator — Maidstone & Tunbridge Wells NHS Trust
Locations (1):
- Maidstone Hospital, Maidstone, Kent, United Kingdom